CLINICAL TRIAL: NCT04701697
Title: Phase Ib Study of Recombinant Human Albumin Injection for the Treatment of Ascites in Patients With Hepatic Cirrhosis
Brief Title: Phase Ib of Recombinant Human Albumin Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-2019-002
Record Dates: First submitted 2020-11-29; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-11

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active comparator：HumanAlbumin (Active Comparator): Participants received HumanAlbumin 10g/d
  Interventions: Drug: HumanAlbumin
- Experimental:Recombinant Human Albumin Injection 10g (Experimental): Participants received Recombinant Human Albumin Injection 10g/d
  Interventions: Drug: Recombinant Human Albumin Injection
- Experimental:Recombinant Human Albumin Injection 20g (Experimental): Participants received Recombinant Human Albumin Injection 20g/d
  Interventions: Drug: Recombinant Human Albumin Injection
- Experimental:Recombinant Human Albumin Injection 30g (Experimental): Participants received Recombinant Human Albumin Injection 30g/d
  Interventions: Drug: Recombinant Human Albumin Injection

INTERVENTIONS:
Drug: Recombinant Human Albumin Injection — Participants will receive Recombinant Human Albumin Injection of intravenous infusion
  Other Names: Intravenous infusion of human albumin injection
  Arms: Experimental:Recombinant Human Albumin Injection 10g; Experimental:Recombinant Human Albumin Injection 20g; Experimental:Recombinant Human Albumin Injection 30g
Drug: HumanAlbumin — Participants will receive HumanAlbumin of intravenous infusion
  Other Names: Intravenous infusion of recombinant human albumin injection
  Arms: active comparator：HumanAlbumin

SUMMARY:
A Randomized, Multicenter,Open-label, positive-controlled, Multi-dose Phase 1 Study to Evaluate the Safety, Tolerance,Efficacy, Pharmacokinetics and Immunogenicity of recombinant human albumin injection in Patients With Hepatic Cirrhosis

DETAILED DESCRIPTION:
This study was to evaluate the safety, tolerability,efficacy, pharmacokinetics and immunogenicity of recombinant human albumin injection in Patients With Hepatic Cirrhosis. The study design consists of two phases: Screening and treatment phase(dose increasing stage).Following the Screening phase, all eligible subjects will be randomized to receive recombinant human albumin injection or HumanAlbumin, study medication in a 3:1 ratio.Dose increasing stage (including 3 dose groups with increasing dose, and each group was set with HumanAlbumin control).The initial dose was 10g. The highest dose group was set at 30g.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age;
2. No less than 45 kg.
3. Diagnosed with ascites due to cirrhosis.

Exclusion Criteria:

1. Allergy to biological products;
2. West-Haven HE ≥ III ;
3. Uncontrolled severe infections;
4. HRS. Serum creatinine (Cr)>2×ULN, or Cr increase>50% during the screening period;
5. Combined with other serious underlying diseases.
6. Organ transplant recipients;
7. Child-bearing females. Pregnancy test positive. Refusing to take contraceptive measures; (8) Participation in other clinical trials. Using study drugs within three month; (9) With the following laboratory test abnormality:

   1. PLT<30×109/L, HGB<70 g/L;
   2. ALT and (or) AST> 5×ULN, TBIL>3×ULN;
   3. Prothrombin activity <40%, PT prolonged>5s;
   4. LVEF <50%;
   5. The 24h urine volume exceeds 1500 mL/day ;

10) Other subjects by investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance | Day 1-Day 14（approximately，After the treatment）
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Major efficacy character: Albumin concentration change | Day 1-Day 14（approximately，After the treatment）
  Albumin concentration change from baseline to Day 14（approximately，After the treatment）
Efficacy：Ascites regression rate | Day 1-Day 14（approximately，After the treatment）
  Ascites regression rate from baseline at Day 14（approximately，After the treatment）
Efficacy：Ascites resolution time | Day 1-Day 14（approximately，After the treatment）
  Ascites resolution time
Efficacy： HRS (hepato-renal syndrom) | Day 1-Day 14（approximately，After the treatment）
  Incidence of HRS
Efficacy： OHE(overt hepatic encephalopathy) | Day 1-Day 14（approximately，After the treatment）
  Incidence of OHE
Efficacy： abdominal circumference | Day 1-Day 14（approximately，After the treatment）
  Change of abdominal circumference from baseline at Day 14（approximately，After the treatment）
Efficacy：Weight | Day 1-Day 14（approximately，After the treatment）
  Change of Weight from baseline at Day 14（approximately，After the treatment）
Pharmacodynamic parameters | Day 1-Day 29
  Plasma colloidal osmotic pressure change from baseline
PK parameters | Day 1-Day 29
  Maximum Plasma Concentration（Cmax）of ALB as Recombinant Human Albumin administration occur
PK parameters | Day 1-Day 29
  Time to Maximum Plasma Concentration（Tmax）of ALB as Recombinant Human Albumin administration occur
PK parameters | Day 1-Day 29
  Half life (t1/2）as Recombinant Human Albumin administration occur
PK parameters | Day 1-Day 29
  Area under the curve(AUC) as Recombinant Human Albumin administration occur
Immunogenicity | Day 1-Day 29
  Percentage of patients with positive reaction against human albumin

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Dr, Study Director — The first affiliated hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Wang X, Li W, Kong F, Guo X, Jin Q, Gao R, Hu Y, Cai Y, Xin G, Ji H, Piao H, Fu Z, Wang Y, Piao Z, Wang S, Hua R, Wen X, Qi Y, Jin J, Wang C, Wang Z, Xu F, Zhou Q, Li X, Yu G, Wang Y, Yang T, Xiang W, Pan Y, Niu J, Gao Y. A randomized, phase Ib trial of recombinant human serum albumin in cirrhotic patients with ascites. Hepatol Int. 2025 Jul 23. doi: 10.1007/s12072-025-10871-x. Online ahead of print. PMID 40699522